CLINICAL TRIAL: NCT06462963
Title: OligoCare TwiCs (Trials Within Cohorts) Trial Comparing Acute Toxicity in Single-fraction vs Multiple-fraction SBRT for Metastasis-directed Treatment (SPRINT)
Acronym: SPRINT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-2387
Record Dates: First submitted 2024-05-28; First posted 2024-06-17 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer; Prostate Cancer; NSCLC; Colorectal Cancer; Oligometastatic Disease
Keywords: radiotherapy; SBRT; TwiCs
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- single-fraction SBRT (Experimental): All lesions to be treated with radical radiotherapy will be treated with single-fraction SBRT, delivered using a dose ranging from 16 Gy to 34 Gy, depending on metastasis location. Acceptable ablative doses are developed in the protocol (see Section 6.4).
  Radiotherapy treatment will last from one single visit to a few weeks, depending on the number of treated metastases.
  Interventions: Radiation: single-fraction SBRT
- multiple-fraction SBRT (Active Comparator): All lesions to be treated with radical radiotherapy will be treated with multiple-fraction SBRT.
  Interventions: Radiation: multiple-fraction SBRT

INTERVENTIONS:
Radiation: single-fraction SBRT — Single-fraction SBRT (Stereotactic Body Radiation Therapy) is a precise form of radiation therapy that delivers a high dose of radiation in a single treatment session to a targeted area, often used for treating small, well-defined tumors. This approach minimizes exposure to surrounding healthy tissues while effectively treating the tumor.
  Arms: single-fraction SBRT
Radiation: multiple-fraction SBRT — Multiple-fraction SBRT (Stereotactic Body Radiation Therapy) is a precise form of radiation therapy that delivers high doses of radiation over several treatment sessions to a targeted area, typically used for treating small, well-defined tumors. This method helps to further protect surrounding healthy tissues by spreading the total radiation dose over multiple sessions.
  Arms: multiple-fraction SBRT

SUMMARY:
The goal of this clinical trial is to evaluate single-fraction metastases-directed SBRT in the broader radiation oncology community and to compare its safety and efficacy profile with the current Standard of Care (SoC) of multiple-fraction SBRT in patients with oligometastatic disease of primary breast, prostate, NSCLC and colorectal cancer having all lesions that will be treated with radical radiotherapy amenable to single-fraction SBRT.

The main question/hypothesis this clinical trial aims to answer is:

- Single-fraction SBRT has comparable outcomes as those obtained with multiple fraction SBRT, both in terms of safety and efficacy.

Patients from the OligoCare cohort will be randomized to receive either single-fraction SBRT or the current SoC of multiple-fraction SBRT.

DETAILED DESCRIPTION:
As a consequence of improved survival of metastatic cancer patients due to more effective systemic therapy, focused radiotherapy in the form of stereotactic body radiotherapy (SBRT) has become a standard of care in many clinical situations to achieve durable symptom and / or metastasis control: treatment of brain metastases, of painful bone or spinal metastases and especially as local treatment in a multimodality treatment strategy for oligometastatic disease. These indications are supported by international practice guidelines, e.g. ESMO guidelines for NSCLC and colorectal cancer; and NCCN guidelines for NSCLC, prostate cancer, renal cell cancer, colorectal cancer and sarcoma.

However, despite the universal use of SBRT in the local treatment of oligometastases, the level of evidence supporting stereotactic radiotherapy is low, apart from few small prospective clinical trials showing a very favourable toxicity profile of SBRT and promising efficacy data. In this context, the OligoCare research project, a prospective observational cohort study, has been developed within the E²-RADIatE platform. The aim of this project is to collect real-world data on SBRT treatment of patients with oligometastatic disease of primary breast, prostate, lung and colorectal cancer, with no limit on the maximum number of treated metastases.

Yet, the local treatment of multiple metastases poses several challenges. One of them is the integration of local metastases-directed SBRT into a systemic treatment strategy: in an interim analysis of the OligoCare cohort, almost all patients were treated with fractionated SBRT and the median number of SBRT fractions was 5. This would result in a total of 50 SBRT fractions in a patient with 10 metastases. Considering that several drugs are paused before and after SBRT, the systemic therapy free interval could last for almost 2 months, which one could consider as unacceptably long in metastatic cancer patients.

One solution to this problem would be the delivery of radiotherapy in a smaller number of SBRT fractions, preferably as single-fraction SBRT. Single-fraction SBRT has been described since the 90's for treatment of liver metastases, lung metastases or vertebral metastases. A recent randomized phase II trial compared multiple-fraction vs single-fraction SBRT for pulmonary oligometastases (n=90) and did not observe differences in toxicity or any oncological outcome parameter.

Nevertheless, single-fraction SBRT still lacks adoption in the radiation oncology community. Likely reasons are the experience of single-fraction SBRT restricted to small, highly specialized centers, the small number of patients treated with single-fraction SBRT in the literature and the concerns of potentially increased toxicity and / or decreased efficacy.

There is consequently a strong rationale to implement and evaluate single-fraction metastases-directed SBRT in the broader radiation oncology community and to compare its safety and efficacy profile with the current SoC of multiple-fraction SBRT.

This question will be addressed in the current Trials within Cohorts (TwiCs) study, in which patients from the OligoCare cohort will be randomized to receive either single-fraction SBRT or the current SoC of multiple-fraction SBRT. The main hypothesis is that single-fraction SBRT has comparable outcomes as those obtained with multiple fraction SBRT, both in terms of safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Patient is part of the RP1822-OligoCare. As in OligoCare, ALL active cancer lesions (loco-regional primary and all oligometastases) were or will be treated with radical intent (surgery or radiotherapy).
* All lesions that will be treated with radical radiotherapy have to be amenable to single-fraction SBRT. Concurrent systemic treatment is allowed.
* Written informed consent must be given according to ICH/GCP, and national/local regulations. Patients will be consented in a step-wise approach.

Step 1 [both control and experimental arms]: patients will need to consent to be included and evaluated in E²-RADIatE (that includes the non-interventional OligoCare prospective registry cohort) and to potentially be randomized to future sub-studies for which they are eligible; no further consent will be sought if they are randomized to the SoC (control) arm; Step 2 [experimental arm only]: if eligible for the current sub-study and randomized to receive single-fraction SBRT, patients will need to consent to receiving the experimental treatment.

Exclusion Criteria:

All targeted lesion judged by the treating physician to be associated with risks for severe toxicity following single-fraction SBRT. The following lesions are systematically excluded:

* Pulmonary metastases within 1 cm of proximal bronchial tree, esophagus or brachial plexus
* Metastases within < 5 mm of any hollow GI structure: esophagus, stomach, small bowel, large bowel
* Metastases within < 5 mm of the spinal cord, the cauda equina or the brachial plexus
* Metastases > 5 cm in largest diameter.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 302 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2029-02-15 (Estimated); Study Completion 2029-02-15 (Estimated)

PRIMARY OUTCOMES:
Grade 3+ SBRT-related toxicity | within 12 months following treatment with radical radiotherapy.
  The cumulative incidence of grade 3+ SBRT-related toxicity within 12 months following treatment with radical radiotherapy. This study will use the International Common Terminology Criteria for Adverse Events (CTCAE), version 5.0, for adverse event reporting.

SECONDARY OUTCOMES:
Progression free survival (PFS) | 4.5 years from first patient in
  defined as the time from the date of randomization to the date of first progression (local, regional or distant) as per local assessment or death.
Overall survival (OS) | 4.5 years from first patient in
  defined as the time from the date of randomization to the date of death from any cause.
Local control (LC) | 4.5 years from first patient in
  defined as freedom from local metastasis (inside the PTV or prior treated field).
Pattern of progression of primary disease and metastases | 4.5 years from first patient in
  Pattern of progression of primary disease and metastases includes local, regional and/or distant progression or recurrence.

OTHER OUTCOMES:
Health-related Quality of life (HRQoL) | 4.5 years from first patient in
  The magnitude of change in HRQoL in terms of physical functioning from EORTC QLQ-C30.
Health-related Quality of life (HRQoL) | 4.5 years from first patient in
  The magnitude of change in HRQoL in terms of pain/discomfort from EQ5D-5L questionnaires.
Economic impact of radiation treatment | 4.5 years from first patient in
  To document the health economic impact of the two treatments by collecting Use of resources questionnaires during radiation treatment and during follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Guckenberger, MD, Principal Investigator — Radiation Oncology, University of Zurich, Switzerland; Piet Ost, MD, Principal Investigator — GZA Sint-Augustinus, Wilrijk, Belgium
Locations (15):
- Belgium (5):
  - Onze Lieve Vrouw Ziekenhuis, Aalst
  - Institut Jules Bordet, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - AZ Groeninge Kortrijk, Kortrijk
  - Ziekenhuis aan de Stroom (ZAS) - ZAS Augustinus, Wilrijk
- Italy (6):
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - Istituto Clinico Humanitas, Milan
  - Istituto Europeo di Oncologia, Milan
  - Sacro Cuore Hospital, Negrar
  - Policlinico Universitario Campus Bio-Medico- Oncology Center, Roma
  - Universita Di Torino, Torino
- Netherlands (2):
  - Radiotherapiegroep Arnhem, Deventer
  - Radboudumc - Radboud University Medical Center Nijmegen, Nijmegen
- Switzerland (2):
  - Inselspital - Inselspital, Bern
  - UniversitaetsSpital Zurich, Zurich